CLINICAL TRIAL: NCT00668512
Title: Phase I Study To Evaluate The Toxicity And Feasibility Of Intratumoral Injection Of Alpha-Gal (Beta-galactosidase ) Glycosphingolipids In Patients With Advanced Melanoma
Brief Title: Intratumoral Injection Of Alpha-Gal Glycosphingolipids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Giles Whalen, Principal Investigator, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UM200701
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Melanoma
Keywords: metastatic cutaneous melanoma; alpha-gal glycolipids
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antimelanoma injection-GSL alpha-Gal (Experimental): Intervention consists of injection of a single melanoma metastasis with two injections of GSL alpha-Gal separated by four weeks. Both injections done with the same dose of GSL alpha-GAL each time. Phase 1 dose escalating scheme: 0.1mg, 1 mg, 10mg
  Interventions: Biological: Antimelanoma injection of GSL alpha-Gal

INTERVENTIONS:
Biological: Antimelanoma injection of GSL alpha-Gal — Single arm, phase 1 trial of escalating doses of GSL alpha-Gal (0.1mg, 1mg, 10mg)injected into a melanoma metastasis at day 0 and then again 4 weeks later.
  Other Names: Alph-Gal Glycosphingolipids

SUMMARY:
This is a Phase I pilot study to evaluate the toxicity of two intra-tumoral injections of GSL alpha-GAL in patients with advanced or metastatic cutaneous melanoma. Patients who have failed standard therapies or are not eligible for standard treatment will be eligible for this study.

DETAILED DESCRIPTION:
A standard Phase I dose escalation model will be used to define the maximum tolerated dose (MTD) of GSL alpha-GAL that can be administered directly into the tumor lesion on two separate injections separated by 4-weeks. This trial will serve as the basis for future Phase II trials utilizing multiple injections of GSL alpha-GAL in refractory solid tumors.

Additionally, in this study we will look for histologic evidence of an immune response against the injected melanoma lesions which matches that seen in mice. Our hypothesis for this study is that a second injection of GSL alpha-GAL into a melanoma lesion will not precipitate an allergic or autoimmune reaction, but will cause a histologically evident immune response to the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent melanoma who have failed standard therapies, or are not candidates for standard therapies.
2. Patients must have at least one measurable cutaneous lesion that is accessible and suitable for injection of the GSL alpha-GAL.
3. Patients should not be undergoing any active treatment with chemotherapy, radiotherapy, or steroids (either because the patient or the treating physician has decided not to employ these therapies at this time, or because they had already been tried and failed). If they have been treated with these modalities, the treatments should have been completed at least two weeks prior to date of injection of GSL alpha-GAL.
4. Patients should be judged by the investigator to be able to undergo safely the procedure needed to inject the tumor with GSL alpha-GAL.
5. Age >18 years old.
6. ECOG (Eastern Cooperative Oncology Group) performance of <2. International Normalized Ratio (INR)<1.5 and a PTT (partial thromboplastin time ) no greater than normal limits within 1 week prior to intra-tumoral injection (For patients who may be on blood thinners)
7. Laboratory Criteria (completed <2 weeks before enrollment) Hematologic: (White Blood Cell Count) WBC > 3500/mm3 or (absolute neutrophil count) ANC > 1500/mm3 and platelet count > 100 000/ mm3 Hepatic: Total bilirubin < 4.0 mg/dl Renal: Creatinine < 2.2 mg/dl.
8. Patients must be negative for HIV (circulating antibody), Hepatitis B (circulatory antigen), and Hepatitis C (circulating antibody).
9. Patients should have an expected survival of >6 weeks and should not have other systemic anti-tumor treatments planned during this time frame.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not eligible:

1. Patients who are pregnant or nursing (PRN serum pregnancy test to be done at week -1).
2. Patients under the age of 18.
3. Patients with severe infections or septicemia.
4. Patients with a history of autoimmune disease.
5. Patients in, or about to be in, active treatment with chemotherapy or steroids.
6. Patients who refuse HIV/hepatitis testing and patients who do not sign an approved consent form
7. Patient has received other investigational drugs within 14 days before enrollment or is expected to participate in an experiment drug study during this study treatment.
8. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Grade 3/4 toxicity | 11-12 weeks
  Grade 3/4 toxicity or adverse event during injection protocol or up to a month after

SECONDARY OUTCOMES:
Clinical response | 2 years
  Injected tumor deposit regression (RECIST), regression of other known metastases (RECIST), progression of disease (new metastases)

OTHER OUTCOMES:
Immune response in injected lesion | six weeks
  Evidence of immune cell infiltration of injected tumor: histologic comparison of biopsy of injected lesion with pre injection biopsy of same lesion

CONTACTS AND LOCATIONS:
Overall Officials: Giles Whalen, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Universiity of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Background] Malmberg KJ. Effective immunotherapy against cancer: a question of overcoming immune suppression and immune escape? Cancer Immunol Immunother. 2004 Oct;53(10):879-92. doi: 10.1007/s00262-004-0577-x. Epub 2004 Jul 28. PMID 15338206
- [Background] Spiotto MT, Fu YX, Schreiber H. Tumor immunity meets autoimmunity: antigen levels and dendritic cell maturation. Curr Opin Immunol. 2003 Dec;15(6):725-30. doi: 10.1016/j.coi.2003.09.018. PMID 14630209
- [Result] Lugade AA, Moran JP, Gerber SA, Rose RC, Frelinger JG, Lord EM. Local radiation therapy of B16 melanoma tumors increases the generation of tumor antigen-specific effector cells that traffic to the tumor. J Immunol. 2005 Jun 15;174(12):7516-23. doi: 10.4049/jimmunol.174.12.7516. PMID 15944250